CLINICAL TRIAL: NCT03116399
Title: PRISM 2.0 in Diverse Living Contexts With Diverse Populations of Older Adults
Brief Title: PRISM 2.0 in Diverse Living Contexts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1811019713; 3P01AG017211 (NIH)
Record Dates: First submitted 2017-03-27; First posted 2017-04-17 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: Social Isolation in Older Adults
Keywords: Older adults; Social Support; Technology uptake

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM 2.0 Condition (Experimental): Exposing participants to the PRISM 2.0 interface.
  Interventions: Behavioral: PRISM 2.0 Condition
- Tablet Condition (Placebo Comparator): Exposing participants to the regular computer/tablet
  Interventions: Behavioral: Tablet Condition

INTERVENTIONS:
Behavioral: PRISM 2.0 Condition — Access to the PRISM 2.0 program
  Arms: PRISM 2.0 Condition
Behavioral: Tablet Condition — Access to the tablet
  Arms: Tablet Condition

SUMMARY:
The focus of the study is to evaluate the expanded version of PRISM 1.0 for a broad array of seniors with different needs and circumstances. The aims of the study are to: 1) obtain information on perceptions of the usefulness and usability of PRISM 2.0 and interface design issues; 2) examine the impact of access to PRISM 2.0 on social connectivity, engagement, social support, and perceived loneliness; 3) examine the impact of access to PRISM 2.0 on perceived isolation, well-being, and quality of life; 4) examine the impact of access PRISM 2.0 on computer attitudes, self-efficacy, technology proficiency and technology uptake; 5) gather data on usefulness of system features and if these vary by living condition; and 6) examine, in our statistical models, the influence of factors such as age, cognitive abilities, ethnicity, education on system use and outcomes.

DETAILED DESCRIPTION:
This study is part of the CREATE center. The focus of the study is to evaluate the expanded version of PRISM 1.0 for a broad array of seniors with different needs and circumstances. The aims of the study are to: 1) obtain information on perceptions of the usefulness and usability of PRISM 2.0 and interface design issues; 2) examine the impact of access to PRISM 2.0 on social connectivity, engagement, social support, and perceived loneliness; 3) examine the impact of access to PRISM 2.0 on perceived isolation, wellbeing, and quality of life; 4) examine the impact of access PRISM 2.0 on computer attitudes, self-efficacy, technology proficiency and technology uptake; 5) gather data on usefulness of system features and if these vary by living condition; and 6) examine, in our statistical models, the influence of factors such as age, cognitive abilities, ethnicity, education on system use and outcomes. The design of the PRISM 2.0 is well grounded and the chosen features will be based on: 1) the findings from the PRISM 1.0 trial; 2) the cognitive, human factors and engineering; 3) emerging findings in aging (e.g., findings related to technology acceptance, social isolation, social networks, life engagement); 4) existing theories of aging (e.g., Stress-Process Model; Active Theory; Social Isolation/Engagement; 5) findings regarding the benefits of technology for seniors; 6) findings from previous work from CREATE regarding interface design, training, provision of environmental support, and the needs of older adults; 7) recent findings regarding Internet use among older adults; 8) findings from our prior focus groups on barriers to access of technology and technology preferences; 9) findings from our technology-based community intervention programs with older adults; 10) existing models of technology adoption and diffusion; 11) the literature on implementation science our planned focus groups and pilot testing of PRISM 2.0.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+ years
* Able to read English at the 6th grade level
* Passing score of Social Isolation Screening
* Passing score of brief Technology Proficiency Screen
* Passing score of Telephone Interview for Cognitive Status (TICS)
* Passing score of Woodcock Johnson Reading Comprehension (Spanish equivalent)
* Passing score of Fuld Object Memory Evaluation

Exclusion Criteria:

* Blind or deaf
* Has terminal Illness or severe motor impairment
* Significant use of computer/Internet/email in the home or elsewhere
* Working for a paid more than 5 hours/week
* Participate as formal volunteer more than 5 hours/week
* Attend senior center or another formal organization for than 10 hours/week

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J. Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Florida State University, Tallahassee, Florida
  - Georgia Institute of Technology, Atlanta, Georgia
  - University of Illinois at Urban-Champagne, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Czaja SJ, Charness N, Rogers WA, Sharit J, Moxley JH, Boot WR. The Benefits of Technology for Engaging Aging Adults: Findings From the PRISM 2.0 Trial. Innov Aging. 2024 Apr 25;8(6):igae042. doi: 10.1093/geroni/igae042. eCollection 2024. PMID 38854853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on response to study recruitment efforts (e.g., flyers, mailings, etc.) at 3 research centers between April 2017 and March 2020.
Period: Overall Study
Arm/Group | PRISM 2.0 Condition | Tablet Condition
Started | 128 | 120
6-month | 98 | 108
9-month | 91 | 101
Completed | 88 | 96
Not Completed | 40 | 24
Not completed — Death | 8 | 3
Not completed — Lost to Follow-up | 7 | 11
Not completed — Investigator Decision | 1 | 1
Not completed — Withdrawal by Subject | 24 | 9

BASELINE CHARACTERISTICS:
Population: We are unable to report baseline for 3 participants in the PRISM 2.0 Condition arm as their data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRISM 2.0 Condition | Tablet Condition | Total
Number analyzed (Participants) | 125 | 120 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 125 | 117 | 242
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76 [71 to 84] | 75 [70 to 84.5] | 76 [70 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants in the PRISM 2.0 Condition did not report this measure.
  Participants
    number analyzed (Participants) | 123 | 120 | 243
    Female | 100 | 89 | 189
    Male | 23 | 31 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 2 | 23
  Not Hispanic or Latino | 100 | 115 | 215
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 20 | 46
  White | 84 | 94 | 178
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 125 | 120 | 245
Functional Health/Well-being as Measured by Modified SF-36, a Self-report Measure [Median (Inter-Quartile Range); unit: units on a scale] — A self-report measure of functional health and well-being ranging from 0 (poor functional health/well-being) to 1400 (better functional health/well-being). Population: 8 participants in the PRISM 2.0 Condition and 5 participants in the Tablet Condition did not have SF-36 data at baseline.
  units on a scale
    number analyzed (Participants) | 117 | 115 | 232
    (all) | 855 [765 to 970] | 865 [785 to 950] | 857.5 [775.2 to 960]
Loneliness as Measured by Loneliness Scale, a 20-item Scale to Measure One's Subjective Feelings [Median (Inter-Quartile Range); unit: units on a scale] — A 20-item scale used to measure one's subjective feelings of loneliness and feelings of social isolation ranging from 0 (low level of loneliness) to 80 (high level of loneliness). Population: 5 participants in the PRISM 2.0 Condition and 2 participants in the Tablet Condition did not report Loneliness data at baseline.
  units on a scale
    number analyzed (Participants) | 120 | 118 | 238
    (all) | 39 [33 to 46] | 39 [33 to 48] | 39 [33 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Health/Well-being as Measured by Modified SF-36, a Self-report Measure of Functional Health and Well-being.
Description: Higher score means better functional health/well-being. A lower score reflects poorer health. Range (0-1400)
Time Frame: Baseline, 6 month follow-up and 9 month follow-up
Population: Eleven participants in the PRISM 2.0 arm and 5 participants in the Tablet arm at baseline, 13 participants in the PRISM 2.0 arm and 14 participants in the Tablet arm at the 6-month time point, and 10 participants in the PRISM 2.0 arm and 11 participants in the Tablet arm at 9-month did not complete this measure.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PRISM 2.0 Condition | Tablet Condition
Number analyzed (Participants) | 117 | 115
units on a scale
  Baseline | 855 [765 to 970] | 865 [785 to 950]
  6-month: number analyzed (Participants) | 85 | 94
  6-month | 900 [775 to 990] | 870 [775 to 970]
  9-month: number analyzed (Participants) | 81 | 90
  9-month | 860 [725 to 960] | 857.5 [775 to 960]

2. Secondary Outcome: Change in Loneliness as Measured by Loneliness Scale, a 20-item Scale to Measure One's Subjective Feelings of Loneliness and Feelings of Social Isolation.
Description: Higher score indicates a greater degree of loneliness. A lower score reflects a lower degree of loneliness. Range (0-80)
Time Frame: Baseline, 6 month follow-up and 9 month follow-up
Population: Data is unavailable for 8 participants in the PRISM 2.0 arm and 2 participants in the Tablet arm at baseline as they did not complete this measure. Missing data is due to normal attrition and special circumstances associated with the COVID-19 pandemic.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PRISM 2.0 Condition | Tablet Condition
Number analyzed (Participants) | 120 | 118
units on a scale
  Baseline | 39 [33 to 46] | 39 [33 to 48]
  6 month: number analyzed (Participants) | 85 | 92
  6 month | 37 [30 to 46] | 36 [31 to 43]
  9 month: number analyzed (Participants) | 77 | 85
  9 month | 35 [29 to 44] | 33 [29 to 41]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PRISM 2.0 Condition | Tablet Condition
All-Cause Mortality (participants affected / at risk) | 8/128 | 3/120
Serious Adverse Events (participants affected / at risk) | 5/128 | 3/120
Other Adverse Events (participants affected / at risk) | 9/128 | 7/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRISM 2.0 Condition (N=128) | Tablet Condition (N=120)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Breast cancer (Reproductive system and breast disorders) | 0 | 1
Heart Conditions (Cardiac disorders) | 2 | 1
Hip Hematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Surgery (Musculoskeletal and connective tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRISM 2.0 Condition (N=128) | Tablet Condition (N=120)
Self-reported depression (Psychiatric disorders) | 7 | 4
Heart Attack (Cardiac disorders) | 0 | 1
Bleeding Ulcer (Gastrointestinal disorders) | 1 | 0
Broken Hand (Musculoskeletal and connective tissue disorders) | 0 | 1
Pacemaker Surgery (Cardiac disorders) | 0 | 1
Spinal problems (Musculoskeletal and connective tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Due to COVID-19, the trial was disrupted as the respect universities and facilitators serving seniors were closed. Thus, the trial protocol needed to be revised resulting in delays in data collection. Further, the "lock-down" resulted in delays in data entry and cleaning as the research personnel were not permitted on their respective campuses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03116399/Prot_SAP_000.pdf